CLINICAL TRIAL: NCT02222883
Title: Prevalence of BRCA in Patients With Primary or Platinum Sensitive Recurrent Ovarian Cancer.
Brief Title: Prevalence of BRCA in Patients With Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: AGO Research GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: AGO-TR 1
Record Dates: First submitted 2014-08-19; First posted 2014-08-21 (Estimated); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: BRCA Status; Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA Blood sample Tumorblock
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients with primary diagnosis: patients with primary diagnosis of ovarian cancer for testing of BRCA status regarding germline and somatic mutation
  Interventions: Genetic: Testing of BRCA status regarding germline and somatic mutation
- patients with platinum-sensitive recurrence: patients with platinum-sensitive recurrence of ovarian cancer for testing of BRCA status regarding germline and somatic mutation
  Interventions: Genetic: Testing of BRCA status regarding germline and somatic mutation

INTERVENTIONS:
Genetic: Testing of BRCA status regarding germline and somatic mutation

SUMMARY:
The aim of this prospective registration and translational research study is to evaluate the praevalence of BRCA regarding germline and somatic mutations.

DETAILED DESCRIPTION:
Explorative analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Female ovarian cancer patients aged >= 18 years.
* Women with first diagnosis of epithelial ovarian cancer OR women diagnosed with platinum-sensitive recurrent ovarian cancer.
* Multiple platinum based prior therapies are allowed.

Exclusion Criteria:

* Non-epithelial ovarian malignancy.
* Platinum-resistant or refractory disease.
* Paraffin embedded tumor samples not available.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 500 consecutive patients (up to 250 patients with primary diagnosis and up to 250 patients with platinum-sensitive recurrence of ovarian cancer.
Sampling Method: Probability Sample
Enrollment: 530 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Germline alterations in BRCA1/2 (yes/no) and other ovarian cancer predisposing genes (yes/no; if yes which) | once per sample

SECONDARY OUTCOMES:
Results of Immunohistochemistry in tumor samples | once per sample
Somatic alterations in BRCA1/2 (yes/no) and other ovarian cancer predisposing genes (yes/no; if yes which) | once per sample
BRCAness tumor phenotype in ovarian cancer (yes/no). | once per sample
Differences of tumor samples from primary and relapsed disease | once per sample for each stage of disease
Patient Survey for perspectives and satisfaction regarding testing and counseling | once after BRCA result is available
  3 questions
Determining the correlation of genetic alterations, cancer treatments, overall survival, progression-free survival and occurrence of new malignancies | once

OTHER OUTCOMES:
Validate the results from Pennington et al. (Pennington et al. Clin Cancer Res 2014) | once
Evaluate predictive value of PARp-1 expression for HRD mutations | once for all samples

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Harter, PhD MD, Study Chair — Kliniken Essen-Mitte, Germany
Locations (20):
- Germany (20):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinik Carl Gustav Carus, Dresden
  - Evangelisches Krankenhaus, Düsseldorf
  - Kliniken Essen-Mitte, Essen
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - NCT Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Zentrum für Gynäkologische Onkologie, Kiel
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Universitätsklinikum Gießen und Marburg, Marburg
  - Klinikum rechts der Isar, München
  - LMU München, Klinik Großhadern, München
  - Sana Klinikum Offenbach, Offenbach
  - Universitäts-Frauenklinik, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Dr. Horst Schmidt Kliniken, Wiesbaden
  - Universitätsklinikum Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schouten PC, Richters L, Vis DJ, Kommoss S, van Dijk E, Ernst C, Kluin RJC, Marme F, Lips EH, Schmidt S, Scheerman E, Prieske K, van Deurzen CHM, Burges A, Ewing-Graham PC, Dietrich D, Jager A, de Gregorio N, Hauke J, du Bois A, Nederlof PM, Wessels LF, Hahnen E, Harter P, Linn SC, Schmutzler RK. Ovarian Cancer-Specific BRCA-like Copy-Number Aberration Classifiers Detect Mutations Associated with Homologous Recombination Deficiency in the AGO-TR1 Trial. Clin Cancer Res. 2021 Dec 1;27(23):6559-6569. doi: 10.1158/1078-0432.CCR-21-1673. Epub 2021 Sep 30. PMID 34593530
- [Derived] Hauke J, Harter P, Ernst C, Burges A, Schmidt S, Reuss A, Borde J, De Gregorio N, Dietrich D, El-Balat A, Kayali M, Gevensleben H, Hilpert F, Altmuller J, Heimbach A, Meier W, Schoemig-Markiefka B, Thiele H, Kimmig R, Nurnberg P, Kast K, Richters L, Sehouli J, Schmutzler RK, Hahnen E. Sensitivity and specificity of loss of heterozygosity analysis for the classification of rare germline variants in BRCA1/2: results of the observational AGO-TR1 study (NCT02222883). J Med Genet. 2022 Mar;59(3):248-252. doi: 10.1136/jmedgenet-2020-107353. Epub 2020 Dec 3. PMID 33273034
- [Derived] Hauke J, Hahnen E, Schneider S, Reuss A, Richters L, Kommoss S, Heimbach A, Marme F, Schmidt S, Prieske K, Gevensleben H, Burges A, Borde J, De Gregorio N, Nurnberg P, El-Balat A, Thiele H, Hilpert F, Altmuller J, Meier W, Dietrich D, Kimmig R, Schoemig-Markiefka B, Kast K, Braicu E, Baumann K, Jackisch C, Park-Simon TW, Ernst C, Hanker L, Pfisterer J, Schnelzer A, du Bois A, Schmutzler RK, Harter P. Deleterious somatic variants in 473 consecutive individuals with ovarian cancer: results of the observational AGO-TR1 study (NCT02222883). J Med Genet. 2019 Sep;56(9):574-580. doi: 10.1136/jmedgenet-2018-105930. Epub 2019 Apr 12. PMID 30979843